CLINICAL TRIAL: NCT07028788
Title: Effectiveness of Virtual Mindfulness Combined With Brief Structured Breathing Training on Perceived Stress, Burnout, Sleep Quality, and Cognitive Function Among Rotating-Shift Nurses: A Randomized Controlled Trial
Brief Title: Virtual Mindfulness and Breathing Training for Stress, Burnout, Sleep, and Cognition in Rotating-Shift Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Shih-Chin (Other)
Responsible Party: Sponsor-Investigator, Chang Shih-Chin, Principal Investigator, School of Nursing, National Defense Medical Center, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSGH-PH_E_114018
Record Dates: First submitted 2025-05-18; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Occupational Burnout; Work-Related Stress; Sleep Disturbance; Cognitive Dysfunction; Shift Work Disorder
Keywords: breathing training; burnout; cognitive function; mindfulness meditation; mobile health; perceived stress; physiological arousal; rotating-shift nurse; sleep quality; virtual reality
MeSH Terms: conditions — Burnout, Professional; Occupational Stress; Parasomnias; Cognitive Dysfunction; Burnout, Psychological; Sleep Initiation and Maintenance Disorders | interventions — Respiration

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of four parallel groups: (1) health education control group, (2) mobile-based mindfulness group, (3) mobile-based mindfulness combined with brief structured breathing group, and (4) virtual reality-assisted mindfulness combined with brief structured breathing group. Each group receives a different non-pharmacologic intervention over an 8-week period. The study follows a parallel assignment model without crossover.
Masking Description: This is an open-label trial. Due to the nature of the behavioral interventions and the use of virtual reality or mobile devices, participants and implementers are aware of the assigned group. However, outcome assessors and data analysts will be blinded to group allocation to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Health Education Control Group(CG) (Other): Participants will receive an 8-week electronic health education handbook covering topics such as healthy eating habits, balanced nutrition, the physiological impact of shift work, sleep schedules for shift workers, the effects of electronic device use on sleep, and identifying sources of stress. The content does not include any components related to mindfulness or breathing exercises.
  Interventions: Other: Health Education Material
- Mobile-based Mindfulness Group (MMG) (Experimental): Participants will be guided through mindfulness exercises using a pre-recorded 360-degree natural environment video accessed via a mobile application. Participants in the intervention groups will engage in an 8-week program, practicing five times per week, with each session lasting 10 minutes.
  Interventions: Behavioral: Mobile-Based Mindfulness
- mobile-based mindfulness combined with brief structured breathing training group (MMBG) (Experimental): Participants will be guided through mindfulness combined with brief structured breathing exercises, using a pre-recorded 360-degree nature video delivered through a mobile application. Participants in the intervention groups will engage in an 8-week program, practicing five times per week, with each session lasting 10 minutes.
  Interventions: Behavioral: Mobile-Based Mindfulness combined with Breathing
- Virtual reality-assisted mindfulness combined with brief structured breathing training group (VMBG) (Experimental): Participants will wear a VR headset and immerse themselves in a natural virtual environment while engaging in mindfulness combined with brief structured breathing exercises. Participants in the intervention groups will engage in an 8-week program, practicing five times per week, with each session lasting 10 minutes.
  Interventions: Behavioral: VR-Based Mindfulness combined with Breathing

INTERVENTIONS:
Other: Health Education Material — Weekly electronic health education handbooks covering nutrition, sleep, shift work, stress awareness, and digital device use.
  Arms: Health Education Control Group(CG)
Behavioral: Mobile-Based Mindfulness — Guided mindfulness practice via mobile app using pre-recorded 360° natural environment video.
  Arms: Mobile-based Mindfulness Group (MMG)
Behavioral: Mobile-Based Mindfulness combined with Breathing — Mindfulness training combined with brief structured breathing exercises via mobile app using 360° nature video.
  Arms: mobile-based mindfulness combined with brief structured breathing training group (MMBG)
Behavioral: VR-Based Mindfulness combined with Breathing — Virtual reality-delivered mindfulness and structured breathing training using immersive 360° natural environment video.
  Arms: Virtual reality-assisted mindfulness combined with brief structured breathing training group (VMBG)

SUMMARY:
This randomized controlled trial aims to evaluate the effectiveness of a mobile- and virtual reality-based mindfulness and breathing intervention on stress, burnout, sleep quality, and cognitive function among Rotating-shift nurses. Participants will be randomly assigned to one of four groups: (1) health education control group, (2) mobile-based mindfulness only, (3) mobile-based mindfulness combined with brief structured breathing, and (4) virtual reality-assisted mindfulness combined with brief structured breathing. The intervention will last for 8 weeks, with participants practicing 5 times per week for 10 minutes per session. Primary outcomes include perceived stress, burnout levels, sleep quality, and cognitive function.

DETAILED DESCRIPTION:
Rotating-shift nurses often experience high levels of chronic stress, occupational burnout, and disrupted sleep patterns, which can negatively affect their cognitive function and well-being. This study aims to investigate the effectiveness of technology-assisted mindfulness and breathing interventions in addressing these issues.

A total of four groups will be included in this randomized controlled trial:

1. Control Group (CG): Participants will receive a weekly electronic health education manual for 8 weeks. Topics include healthy eating habits, balanced nutrition, the physiological impact of shift work, sleep hygiene for shift workers, the effects of electronic devices on sleep, and identifying sources of stress. No mindfulness or breathing content is included.
2. Mobile-based Mindfulness Group (MMG): Participants will engage in guided mindfulness practice via a smartphone application, using a pre-recorded 360-degree nature video.
3. Mobile-based Mindfulness with Breathing Group (MMBG): Participants will follow a similar protocol as MMG, with the addition of brief structured breathing exercises embedded in the training.
4. Virtual Reality-based Mindfulness with Breathing Group (VMBG): Participants will wear a VR headset and immerse themselves in a virtual nature setting while engaging in combined mindfulness and structured breathing training. All intervention groups will complete 10-minute sessions, five times per week, for a total of eight weeks.

Primary outcome measures include: Perceived stress (Perceived Stress Scale, PSS-10-C), Occupational burnout (Nursing Burnout Scale), Sleep quality (Pittsburgh Sleep Quality Index, PSQI) and Cognitive function (including attention and memory tasks). Assessments will be conducted at baseline, immediately post-intervention, and at follow-up. This study will provide insights into the comparative effectiveness of mobile and immersive digital interventions for improving mental health and physiological functioning in Rotating-shift nurses.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 and 65 years.
2. Able to understand spoken or written Mandarin or Taiwanese.
3. Employed full-time for at least 3 months with a signed employment contract.
4. Has worked rotating shifts (including day, evening, and/or night shifts) in the past 3 months.
5. Willing to participate and sign informed consent.
6. Registered nurse.
7. A perceived stress score greater than or equal to 50 based on a standardized scale.

Exclusion Criteria:

1. Pregnant or breastfeeding individuals.
2. History of substance abuse (e.g., tobacco, illicit drugs).
3. Alcohol consumption ≥350 ml/week with alcohol content ≥3.5%.
4. Diagnosed or suspected autonomic nervous system disorders.
5. History of severe or unstable cardiovascular disease, cerebrovascular disease, cancer, or end-stage organ failure within the past 6 months.
6. Current diagnosis of psychiatric disorders (e.g., major depressive disorder, schizophrenia), or use of psychiatric or sleep medications (e.g., antidepressants, sedatives).
7. Reported discomfort (e.g., dizziness, nausea) when using virtual reality devices.
8. Engaged in other regular exercise programs, light therapy, or mind-body interventions during the study period.
9. Participating in other clinical trials simultaneously.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Chinese version of the 10-item Perceived Stress Scale (PSS-10-C ) | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up)
  This scale assesses how unpredictable, uncontrollable, and overloaded individuals perceive their lives to be. It contains two subscales: perceived helplessness and perceived self-efficacy. Each item is rated on a 5-point Likert scale from 0 (never) to 4 (very often). The scale has demonstrated high internal consistency (Cronbach's α = 0.85) and good test-retest reliability (r = 0.66, p < 0.001) over three months in Chinese-speaking nursing samples.
Perceived Stress -Safety Culture Subscale. | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up)
  This measure uses the "Perception of Stress" subscale from the Taiwan version of the Safety Attitudes Questionnaire (SAQ), which includes four items that assess healthcare professionals' awareness of stress and its effects on performance. One item is reverse-coded. Items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Subscale scores are transformed to a 0-100 scale using the formula: Transformed score = (mean score - 1) × 25. Higher scores indicate greater perceived stress. This transformation supports standardization and enables comparison across domains.
Nursing Burnout Scale (NBS) | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up)
  This scale was developed for clinical nurses and evaluates emotional exhaustion, reduced personal accomplishment, and depersonalization. It includes 12 items across three subscales, with four items per subscale. Each item is rated on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The total scale has demonstrated high internal consistency (Cronbach's α = 0.92) and acceptable subscale reliability (Cronbach's α = 0.64-0.86), indicating good psychometric properties for use among nursing professionals.

SECONDARY OUTCOMES:
Actigraphy-Based Sleep Quality Index | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up).
  A composite sleep quality score derived from multiple actigraphy-based parameters including total sleep time, sleep efficiency, number of awakenings, and sleep onset latency. Each parameter will be normalized and weighted based on validated sleep scoring algorithms (e.g., Sadeh algorithm), and then aggregated into a composite index to represent overall sleep quality. Higher scores indicate better sleep.
Sleep quality. Taiwanese version of the Pittsburgh Sleep Quality Index (PSQI-TC ) | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up)
  This outcome measure uses the Taiwanese version of the Pittsburgh Sleep Quality Index (PSQI-TC) to evaluate participants' sleep quality. The PSQI-TC includes 19 items across seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each item is scored from 0 to 3, and total scores range from 0 to 21, with higher scores indicating poorer sleep quality. The scale has demonstrated strong internal consistency, with Cronbach's α ranging from 0.83 to 0.85, and is culturally adapted for use among shift-working nurses in Taiwan.
Cognitive Function - Visual Pursuit Test (VTS-LVT) | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up).
  This test evaluates visual orientation performance and spatial scanning ability under time pressure. The outcome will include accuracy rate and average reaction time (in milliseconds).
Cognitive Function - Determination Test (VTS-DT) | Data will be collected at baseline, 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up).
  This test assesses reactive stress tolerance and decision-making performance under time constraints. The outcome measures include number of errors and average reaction time (in milliseconds).
Cognitive Function - Signal Detection Test (VTS-SDT) | Data will be collected at baseline, 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up).
  This test measures sustained attention and the ability to distinguish relevant signals from distractors. Key outcome variables include hit rate, false alarm rate, and attentional stability.
Heart Rate Variability (HRV) Measured via BVP using Thought Technology System | Baseline (Week 0), Week 4, Week 8, Week 12
  Heart rate variability (HRV) will be measured non-invasively using the Blood Volume Pulse (BVP) sensor of the Thought Technology system (ProComp Infiniti hardware and BioGraph Infiniti software). HRV data will be collected using photoplethysmography (PPG), and derived from inter-beat intervals (IBI). Analysis will include both time-domain indices (e.g., SDNN, RMSSD) and frequency-domain indices (e.g., LF, HF, LF/HF ratio). The assessment will be conducted in accordance with international standards for HRV evaluation and will reflect both sympathetic and parasympathetic autonomic activity. Participants will undergo HRV assessment at Weeks 0 (baseline), 4, 8, and 12 as part of their stress and recovery evaluation.

OTHER OUTCOMES:
Blood Pressure Monitoring Device - Omron HEM-907XL | Data will be collected at baseline (pre-intervention), 4 weeks, 8 weeks (post-intervention), and 12 weeks (follow-up)
  This outcome will include measurements of systolic and diastolic blood pressure using the Omron HEM-907XL, a validated automatic digital sphygmomanometer. Blood pressure will be recorded using the three-reading average method while participants are in a seated resting position. Data will be used for subsequent analysis of cardiovascular responses to intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hui Lin, Ph.D., Study Director — School of Nursing, National Defense Medical Center